CLINICAL TRIAL: NCT00117039
Title: SYNCHRONICITY: A Study to Evaluate the Effectiveness of Aranesp® at 300 Mcg Q3W on Clinical Outcomes in Cancer Patients With Anemia Due to Chemotherapy
Brief Title: A Study to Evaluate the Effectiveness of Aranesp® for Cancer Patients With Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030206
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-08

CONDITIONS: Anemia; Neoplasms
Keywords: anemia; fatigue; Aranesp®; clinical trial
MeSH Terms: conditions — Anemia; Neoplasms; Fatigue | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Aranesp®

SUMMARY:
The purpose of this trial is to assess the effectiveness of Aranesp® administered at 300 mcg every 3 weeks (q3w) in achieving therapeutic objectives of anemia treatment (achieving and maintaining hemoglobin levels consistent with the National Comprehensive Cancer Network (NCCN) guidelines).

ELIGIBILITY:
Inclusion Criteria: - Subjects with non-myeloid malignancy - Anemia (Hgb less than 11.0 g/dL) due to cancer chemotherapy - Receiving chemotherapy and expected to receive at least 8 additional weeks of chemotherapy - Adequate renal function - Adequate liver function Exclusion Criteria: - Subjects with acute myelogenous leukemia (AML), chronic myelogenous leukemia (CML), or myelodysplastic syndromes (MDS) - Unstable cardiac disease - Active bleeding - Active systemic or chronic infection - Severe active chronic inflammatory disease - Other hematologic disorder associated with anemia - Uncontrolled hypertension - Known iron or nutritional deficiency - Known positive test for human immunodeficiency virus (HIV) infection - History of pure red cell aplasia - History of positive antibody response to any erythropoietic agent - Erythropoietin therapy within 4 weeks before screening - RBC transfusions within 2 weeks prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2004-01; Study Completion 2005-04

PRIMARY OUTCOMES:
Hemoglobin maintenance

SECONDARY OUTCOMES:
Quality of Life
Changes in measures of work productivity and anemia treatment convenience

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Boccia R, Lillie T, Tomita D, Balducci L. The effectiveness of darbepoetin alfa administered every 3 weeks on hematologic outcomes and quality of life in older patients with chemotherapy-induced anemia. Oncologist. 2007 May;12(5):584-93. doi: 10.1634/theoncologist.12-5-584. PMID 17522247
- [Result] Boccia R, Malik IA, Raja V, Kahanic S, Liu R, Lillie T, Tomita D, Clowney B, Silberstein P. Darbepoetin alfa administered every three weeks is effective for the treatment of chemotherapy-induced anemia. Oncologist. 2006 Apr;11(4):409-17. doi: 10.1634/theoncologist.11-4-409. PMID 16614237
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/